CLINICAL TRIAL: NCT02731144
Title: The Impact of Optimized Caloric-proteic Nutrition on Clinical Outcome and Physical Component Summary (PCS) of Quality of Life in Septic and Septic Shock Patients
Brief Title: Optimized Caloric-proteic Nutrition in Septic and Septic Shock Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The protocol was modified substantially and will be resubmitted to Clinical Trial
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, MD, PhD, Hospital Sao Domingos
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CEP-HSD 33/2016
Record Dates: First submitted 2016-03-31; First posted 2016-04-07 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2018-01

CONDITIONS: Sepsis; Septic Shock
Keywords: Loss of Physical Function
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental): Individualization of caloric administration with indirect calorimetry and 2.0 to 2.2 g/kg/day of protein. Early initiation of nutritional support (24 hours of admission)
  Interventions: Other: Peptamen intense
- Control group (Active Comparator): Nutritional support initiated in the first 24 hours of admission. Protein and caloric goals calculated as 25 Kcal/kg/day and 1.4 to 1.5 g/kg/day of protein.
  Interventions: Other: Novasource senior

INTERVENTIONS:
Other: Peptamen intense
  Arms: Study group
Other: Novasource senior
  Arms: Control group

SUMMARY:
In this pilot randomized prospective controlled trial the investigators intend to compare the use of a nutritional therapy based on caloric intake determined by indirect calorimetry and high protein intake with nutritional regimen based on 25 Kcal / kg / day and protein intake usually recommended for critically ill patients (1.4 to 1.5 grams / kg / day of protein).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU with sepsis and septic shock according to 3rd International Sepsis Consensus Conference Definitions for sepsis and septic shock
* Mechanically ventilated
* Expected length of stay in ICU ≥ 4 days
* Written informed consent obtained from authorized surrogates

Exclusion Criteria:

* Pregnancy
* Requirement for inspired oxygen content (FIO2) > 0.60
* High output bronchopleural fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Physical function measured through the tool Physical Component Summary - PCS of Short Form 36 | Three months after randomization

SECONDARY OUTCOMES:
Hospital mortality | Up to 1 year
Length of ICU stay | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: JOSE R AZEVEDO, PhD, Principal Investigator — COORDINATOR ICU HOSPITAL SAO DOMINGOS

IPD SHARING:
Plan to Share IPD: Yes